CLINICAL TRIAL: NCT00430937
Title: A Multicenter, Randomized, Assessor-Blind Study to Evaluate Efficacy and Safety of Daptomycin Versus Vancomycin or Teicoplanin for Treatment of Complicated Skin and Soft Tissue Infections (cSSTI)
Brief Title: Efficacy and Safety of Daptomycin Versus Vancomycin or Teicoplanin for Treatment of Complicated Skin and Soft Tissue Infections
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCBC134A2402
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Results first posted 2011-01-05 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Skin Diseases, Infectious; Soft Tissue Infections
Keywords: Complicated Skin and Soft Tissue Infections. Daptomycin, Vancomycin, Teicoplanin; Complicated skin and soft tissue infections
MeSH Terms: conditions — Skin Diseases, Infectious; Soft Tissue Infections | interventions — Daptomycin; Vancomycin; Teicoplanin

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Daptomycin (Experimental): 4 mg/kg intravenous (i.v.) once daily
  Interventions: Drug: Daptomycin
- Pooled Comparator (Active Comparator)
  Interventions: Drug: Vancomycin; Drug: Teicoplanin

INTERVENTIONS:
Drug: Daptomycin — 4 mg/kg intravenous once daily
  Other Names: Cubicin
  Arms: Daptomycin
Drug: Vancomycin — 1 g intravenous twice daily
  Other Names: Vancocin
  Arms: Pooled Comparator
Drug: Teicoplanin — 400 mg intravenous once daily following a loading dose of 400 mg administered at 0, 12, 24 hours on day one.
  Other Names: Targocid
  Arms: Pooled Comparator

SUMMARY:
This study evaluated the efficacy and safety of daptomycin compared to vancomycin or teicoplanin for the treatment of complicated skin and soft tissue infections

ELIGIBILITY:
Inclusion criteria:

* Subjects with a diagnosis of cSSTI
* Infection known or suspected (based on Gram's stain) to be due, at least partially, to Gram-positive bacteria.
* Hospitalised subjects with clinical evidence of at least one of the following:I infected ulcers , major abscess. deep or extensive cellulitis, post-surgical / post-traumatic wound infection
* Presence of at least two of the following: drainage and/or discharge from the infection site, redness, swelling and/or hardened skin, heat and/or localised warmth, pain and/or tenderness to touch, presence of pus.

Exclusion criteria:

* cSSTIs of the following categories:

  * Infected burns,
  * Severely impaired arterial blood supply (such that the likelihood of amputation of the infected anatomical site is likely),
  * Decubitus ulcers,
  * Infected diabetic foot ulcers associated with osteomyelitis,
  * Infected human or animal bites, superficial infections or abscesses in an anatomic site, such as the rectal area, where the risk of anaerobic or Gram-negative pathogen involvement is high (e.g. perirectal abscess),
  * Necrotising fasciitis or gangrene,
  * cSSTI expected to require more than 14 days of intravenous antimicrobial therapy,
  * Skin and/or skin structure infection that can be treated by surgery alone,
  * Infections associated with a permanent prosthetic device that will not be removed within 2 days of study randomisation
* Subjects with documented bacteraemia at Baseline or those with shock or hypotension
* Concomitant clinically suspected or confirmed other site of infection or disorder at study entry that may interfere with the evaluations in this protocol
* Treatment with vancomycin or teicoplanin within the past 48 hours, unless administered for less than 24 hours.
* Subjects admitted to the hospital for conditions associated with rhabdomyolysis or those with an infection due to an organism known prior to study entry to be resistant to daptomycin, vancomycin or teicoplanin.
* Previously diagnosed disease of immune function. Human Immunodeficiency Virus (HIV) infected subjects without Acquired Immune Deficiency Syndrome (AIDS) may be enrolled.
* Subjects receiving oral steroids or receiving immunosuppressant drugs after organ transplant.
* Absence of purulent material for initial culture and Gram's stain. Subjects with cellulitis may be enrolled in the absence of purulent material, provided that infection with a Gram-positive organism is suspected.
* Subjects who have received more than 48 hours of any systemic antibiotic or topical antibiotic at the infection site with activity against Gram-positive pathogens, unless there is clinical evidence of treatment failure OR documented resistance in the identified Gram-positive pathogen to the previous antibiotic therapy.
* cSSTI suspected or documented as being due exclusively to Gram-negative or anaerobic organisms based on epidemiology or on direct examination of a Gram-stained specimen.
* Subjects diagnosed with pneumonia or those with severe renal impairment or hepatic disease
* Previous history of hearing loss. Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2006-04; Primary Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 194 participants were randomized; 5 participants were not exposed to study drug by mistake; therefore, only 189 participants received study drug.
Groups:
- Daptomycin: Daptomycin 4 mg/kg intravenous (i.v.) once daily
- Pooled Comparator: Vancomycin 1 g intravenous (i.v.) twice daily or Teicoplanin 400 mg i.v. once daily following a loading dose of 400 mg administered at 0, 12 and 24 hours on day one.
Period: Overall Study
Arm/Group | Daptomycin | Pooled Comparator
Started | 97 (Additional 5 participants were randomized; however, they were not exposed to study drug by mistake.) | 92
Completed | 70 | 64
Not Completed | 27 | 28
Not completed — Adverse Event | 3 | 8
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 6 | 6
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Protocol Violation | 3 | 2
Not completed — Lack of Efficacy | 6 | 5
Not completed — Inappropriate enrollment | 2 | 1
Not completed — Administrative reasons | 1 | 0
Not completed — Protocol discontinuation criteria met | 1 | 2
Not completed — Unable to classify | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daptomycin | Pooled Comparator | Total
Number analyzed (Participants) | 97 | 92 | 189
Age, Customized [Number; unit: Participants]
  < 65 years | 62 | 61 | 123
  >=65 years | 35 | 31 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 41 | 77
  Male | 61 | 51 | 112

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success as Measured by Comparing the Participants Signs and Symptoms at the "Test of Cure" (TOC) Visit to Those Recorded at Study Baseline in the Clinically Evaluable Population.
Description: Success: Total resolution of clinically significant signs and symptoms of the infection site (cure) or improvement to such a level that no further antibacterial therapy was required (improvement).
  Failure: Persistence or progression of signs and symptoms after at least 3 days of study therapy, or development of new signs and symptoms at the infection site, or concomitant or additional antibacterial therapy with documented activity against isolated organisms, or a treatment duration greater than 14 days, or requirement of a major surgical procedure as adjunct or follow-up therapy.
Time Frame: Baseline to TOC Visit (7-14 days after end of treatment) up to 4 weeks
Population: The clinically evaluable population was used for the efficacy analysis. It included all patients who met the criteria for cSSTI as listed in the Protocol, had no substantive protocol deviation, had a sponsor clinical response assessment of "success" or "failure" at the assessment visit, and had a specified baseline primary site of infection.
Measure: Number; unit: Participants
Arm/Group | Daptomycin | Pooled Comparator
Number analyzed (Participants) | 58 | 47
Participants
  Clinical Success | 53 | 41
  Clinical Failure | 5 | 6

2. Secondary Outcome: Microbiological Efficacy Measured by the Number of Participants Achieving Bacteriological Eradication of Gram-positive Baseline Pathogens at the TOC Visit.
Description: Microbiological Success: All infecting Gram-positive pathogens isolated at baseline were eradicated at the TOC evaluation and a superinfecting pathogen was not isolated either prior to or at the TOC evaluation.
  Microbiological Failure: Persistence of one or more infecting Gram-positive pathogens or isolation of a superinfecting pathogen prior to or at the TOC evaluation.
Time Frame: Baseline to TOC Visit (7-14 days after end of treatment) up to 4 weeks
Population: Population analyzed consisted of patients from the clinically evaluable population who had microbiological assessments.
Measure: Number; unit: Participants
Arm/Group | Daptomycin | Pooled Comparator
Number analyzed (Participants) | 57 | 43
Participants
  Microbiological Success | 56 | 39
  Microbiological Failure | 1 | 4

ADVERSE EVENTS:
Arm/Group | Daptomycin | Pooled Comparator
Serious Adverse Events (participants affected / at risk) | 17/97 | 16/92
Other Adverse Events (participants affected / at risk) | 26/97 | 25/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daptomycin (N=97) | Pooled Comparator (N=92)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Crohn's Disease (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Impaired Healing (General disorders) | 0 | 1
Induration (General disorders) | 1 | 0
Abscess Limb (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 2 | 0
Haemophilus Bacteraemia (Infections and infestations) | 1 | 0
Necrotising Fasciitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Staphylococcal Skin Infection (Infections and infestations) | 1 | 0
Open Wound (Injury, poisoning and procedural complications) | 0 | 1
Creatinine Renal Clearance Decreased (Investigations) | 1 | 0
Diabetic Foot (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemorrhage Intracranial (Nervous system disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Acquired Hydrocele (Reproductive system and breast disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 2
Eczema Nummular (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Graft (Surgical and medical procedures) | 0 | 1
Arterial Occlusive Disease (Vascular disorders) | 2 | 0
Femoral Artery Occlusion (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daptomycin (N=97) | Pooled Comparator (N=92)
Constipation (Gastrointestinal disorders) | 8 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 5 | 5
Alanine Aminotransferase Increased (Investigations) | 2 | 7
Aspartate Aminotransferase Increased (Investigations) | 1 | 5
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 5
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 5
Blood Pressure Increased (Investigations) | 0 | 6
Blood Urea Increased (Investigations) | 1 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 5
Insomnia (Psychiatric disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.